CLINICAL TRIAL: NCT01231542
Title: Phase 1, Open Label, Two Arm, Fixed Sequence Study to Evaluate the Effect of Rifampin and Rifabutin on GSK1349572 Pharmacokinetics in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113099
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1349572; pharmacokinetics; dolutegravir; integrase; rifabutin; rifampin
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Rifampin; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow-up visit 7-14 days after the last dose of study drug. Subjects enrolled in Arm 1 will receive GSK1349572 50 mg once daily for 7 days, GSK1348572 50 mg twice daily for 7 days, and GSK1349572 50 mg twice daily in combination with rifampin 600 mg once daily for 14 days.
  Interventions: Drug: GSK1349572; Drug: Rifampin
- Arm 2 (Experimental): Subjects will have a screening visit within 30 days prior to the first dose of study drug, two treatment periods, and a follow-up visit 7-14 days after the last dose of study drug. Subjects in Arm 2 will receive GSK1349572 50 mg once daily for 7 days and GSK1349572 50 mg once daily in combination with rifabutin 300 mg once daily for 14 days.
  Interventions: Drug: GSK1349572; Drug: Rifabutin

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 is an experimental drug for the treatment of HIV. GSK1349572 is in the integrase inhibitor class. It is not yet approved by the FDA.
Drug: Rifampin — Rifampin is approved by the FDA for the treatment of tuberculosis.
  Other Names: RIFADIN. RIFADIN is a trademark of Sanofi-Aventis
  Arms: Arm 1
Drug: Rifabutin — Rifabutin is approved by the FDA for the treatment of tuberculosis.
  Other Names: MYCOBUTIN. MYCOBUTIN is a trademark of Pfizer
  Arms: Arm 2

SUMMARY:
This study will be a phase I, open label, two arm, fixed sequence crossover study to investigate the effect of rifampin and rifabutin on the steady state pharmacokinetics (PK) of GSK1349572 and the safety and tolerability of GSK1349572 and rifamycin co-administration. Subjects enrolled in Arm 1 will receive GSK1349572 50 mg once daily for 7 days, GSK1348572 50 mg twice daily for 7 days, and GSK1349572 50 mg twice daily in combination with rifampin 600 mg once daily for 14 days. Subjects in Arm 2 will receive GSK1349572 50 mg once daily for 7 days and GSK1349572 50 mg once daily in combination with rifabutin 300 mg once daily for 14 days. Serial PK sampling will be completed following the last dose of each treatment. Safety and tolerability will be assessed throughout the study through assessment of adverse events (AEs), and clinical laboratory tests.

This study will be conducted at one center in the US with healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECG).
* Within 28 or fewer days prior to enrollment, a complete blood count with differential, comprehensive serum chemistry profile, human immunodeficiency virus (HIV) antibody test, and Hepatitis C antibody test will be performed, with the following laboratory values:
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than or equal to upper limit of normal (ULN)
* Hemoglobin greater than or equal to 12.0 for men, greater than or equal to11.0 for women
* Serum creatinine less than or equal to1.5 mg/dL
* Platelet count greater than or equal to 125,000 /cu mm
* Absolute neutrophil count greater than or equal to 1250 /cu mm
* HIV antibody test negative
* Hepatitis C antibody negative
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. or Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for the time period between screening and dosing of study drugs to sufficiently minimize the risk of pregnancy at that point. Female subjects must also agree to use contraception throughout the study and until two weeks after the last dose of study medications.
* Body weight in the range 53-100 kg (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days or 5 half-lives (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks/week for men or >7 drinks/week for women.
* Any illicit drug use within the preceding 2 months.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases.
* History of severe or serious psychiatric disease ever requiring hospitalization, history of suicidal ideation or suicidal attempt, or undergoing psychiatric treatment.
* Site investigator suspicion of active tuberculosis (TB).
* History of Gilbert's disease.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Steady state plasma GSK1349572 concentration at the end of the dosing interval (Cτ) | 28 days
maximum concentration (Cmax) | 28 days
area under the time-concentration curve over the dosing interval (AUC(0-τ)) | 28 days
AUC for a 24-hour interval (AUC(0-24) | 28 days

SECONDARY OUTCOMES:
Subjects with grade 2 or higher adverse events | 28 days
Steady state plasma GSK1349572 minimum plasma concentration (Cmin) | 28 days
time of minimum concentration (tmin) | 28 days
pre-dose concentration (C0) | 28 days
time of maximum concentration (tmax) | 28 days
apparent terminal half-life (t1/2) | 28 days
apparent oral clearance (CL/F) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kawuma AN, Wasmann RE, Dooley KE, Boffito M, Maartens G, Denti P. Population Pharmacokinetic Model and Alternative Dosing Regimens for Dolutegravir Coadministered with Rifampicin. Antimicrob Agents Chemother. 2022 Jun 21;66(6):e0021522. doi: 10.1128/aac.00215-22. Epub 2022 May 23. PMID 35604212